CLINICAL TRIAL: NCT03844022
Title: MRI in McArdle Disease (Glycogen Storage Disease Type V)
Brief Title: MRI in McArdle Disease (GSDV)
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Nicoline Løkken, MD, Research fellow, Rigshospitalet, Denmark
Other Study IDs: H-18023049.1
Record Dates: First submitted 2018-12-12; First posted 2019-02-18 (Actual); Last update posted 2023-02-13 (Actual); Status verified 2023-02

CONDITIONS: Glycogen Storage Disease Type V
MeSH Terms: conditions — Glycogen Storage Disease Type V

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- McArdle disease: Glycogen storage disease
  Interventions: Diagnostic Test: MRI
- Healty controls: Age and gender matched
  Interventions: Diagnostic Test: MRI

INTERVENTIONS:
Diagnostic Test: MRI — magnetic resonance imaging

SUMMARY:
The aim of this study is to describe the degree of muscle wasting in patients with McArdle disease judged by MRI, quantitative magnetic resonance (DIXON) and T1 weighted images, and muscle strength, collected across multiple European sites and compared to healthy controls.

ELIGIBILITY:
Inclusion Criteria:

* GSDV or healthy controls

Exclusion Criteria:

* MRI contradictions

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: McArdle disease (GSDV) Healthy controls
Sampling Method: Non-Probability Sample
Enrollment: 87 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2021-02-01 (Actual)

PRIMARY OUTCOMES:
DIXON MRI | 1 time
  Whole body quantitative muscle fat fraction analyses (DIXON)

SECONDARY OUTCOMES:
Muscle strength | 1 time
  MRC scale
T1 MRI | 1 time
  Whole body qualitative muscle fat fraction analyses (T1)
Back pain questionnaire | 1 time
  Back pain questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Copenhagen Neuromuscular Center, Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No